CLINICAL TRIAL: NCT01922453
Title: Use of Music and Sounds for the External Cephalic Version of Breech Fetuses Near Term.
Brief Title: Music and Sounds for ECV
Acronym: RITMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ritmo-HMO-CTIL
Record Dates: First submitted 2013-08-11; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Breech Presentation; Vertex Presentation
Keywords: breech presentation; vertex presentation
MeSH Terms: conditions — Breech Presentation | interventions — Sound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music and Sound (Experimental): Music and Sound applied to maternal abdomen through a special device for pregnant women.
  Interventions: Other: Music and Sound
- no music and sound (No Intervention)

INTERVENTIONS:
Other: Music and Sound
  Arms: Music and Sound

SUMMARY:
This international study is looking to see if the addition of music and sound on the maternal abdomen encourages fetal position change from breech to vertex in near term women.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women near term with breech presentation.

Exclusion Criteria:

* women with a contraindication for vaginal birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
vertex position | 3 days post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hagit Daum, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel